CLINICAL TRIAL: NCT06313710
Title: Head Down Position for Successful Recanalization of Anterior Circulation Large Vessel Occlusion (HOPES3): a Prospective, Randomized, Open Label, Blinded-end Point, Single-center Study
Brief Title: Head Down Position for Successful Recanalization of Anterior Circulation Large Vessel Occlusion (HOPES4)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2024) 058
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention)
- low dose of head down position (Experimental): -10° Trendelenburg for 30 min
  Interventions: Other: head down position
- high dose of head down position (Experimental): -10° Trendelenburg for 60 min
  Interventions: Other: head down position

INTERVENTIONS:
Other: head down position — -10° Trendelenburg
  Arms: high dose of head down position; low dose of head down position

SUMMARY:
This is a prospective, randomized, open label, blinded-end point, single-center study, aiming to investigate the effect of head down position in anterior circulation large vessel occlusion patients with successful recanalization after endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Anterior circulation large vessel occlusion who received endovascular treatment within 24 hours of stroke onset;
* National Institute of Health Stroke Scale (NIHSS) ≥ 6 before endovascular treatment;
* Successful recanalization (mTICI 2b-3) after endovascular treatment;
* Cerebral circulation time based on DSA of the stroke side was slower than that of the healthy side after successful recanalization;
* ASPECTS ≥ 6 on CT or DWI;
* Absence of parenchymal hematoma on CT images done in the angio suite immediately after the procedure;
* Modified Rankin Scale score before stroke onset ≤ 1;
* Signed informed consent by patient or their legally authorized representative.

Exclusion Criteria:

* Hemorrhagic stroke: cerebral hemorrhage, subarachnoid hemorrhage;
* Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
* After recanalization, severe and sustained (i.e., > 5 minutes) uncontrolled hypertension (systolic blood pressure over 180mmHg or diastolic blood pressure over 105 mmHg) refractory to antihypertensive medication;
* More than four retrieval attempts in the same vessel;
* Cardiac insufficiency (NYHA Class ≥II);
* Pregnancy, plan to get pregnant or during lactation;
* The estimated life expectancy is less than 6 months due to other serious diseases;
* Other conditions unsuitable for this clinical study assessed by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Changes in National Institute of Health stroke scale (NIHSS) | 24±8 hours
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome.

SECONDARY OUTCOMES:
proportion of excellent functional outcome | 90±7 days
  excellent functional outcome is defined as modified Rankin Score (mRS) 0-1. The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
proportion of favorable functional outcome | 90±7 days
  favorable functional outcome defined as modified Rankin Score (mRS) 0-2. The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
ordinal distribution of modified Rankin Score (mRS) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
early neurological improvement (ENI) | 24±8 hours
  ENI is defined as more than 8-point decrease in NIHSS or 0 NIHSS within 24±8 hours
changes in infarct volume | 24±8 hours
  infarct volume is measured by diffused weighted imaging
changes in cerebral edema | 24±8 hours
  cerebral edema is determined by brain imaging
Changes in National Institute of Health stroke scale (NIHSS) | 10±2 days
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome.
new stroke or other vascular event(s) | 90±7 days
proportion of sympomatic intracranial hemorrhage | 24±8 hours
  sympomatic intracranial hemorrhage is defined as a NIHSS increase ≥4 caused by intracranial hemorrhage
proportion of intraparenchymal hemorrhage (PH) | 24±8 hours
  PH was defined as confluent bleeding occupying and causing mass effect
percentage of severe adverse events | 24±8 hours
all-cause mortality | 90±7 days

OTHER OUTCOMES:
changes in dynamic cerebral autoregulation (dCA) | 24±8 hours
  dCA data include phase difference (the main parameter, determined as the phase shift angle ranging from 0° to 90°), gain (difference in the amplitude between CBFV and ABP), and the coherence function (indicates signal-to-noise ratio), which is determined according to previous report (Guo ZN, Guo WT, Liu J, et al. Changes in cerebral autoregulation and blood biomarkers after remote ischemic preconditioning.)
changes in cortical oxygen saturation | 24±8 hours
  cortical oxygen saturation is determined by near infrared spectroscopy
changes in serum biomarkers | 24±8 hours
  serum biomarkers include MMP-9, TNF-alpha, IL-1beta, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Undecided